CLINICAL TRIAL: NCT04896957
Title: Perceptions and Representations of Vaccination Against COVID-19
Acronym: PERCECOVAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Centre Hospitalier Intercommunal Villeneuve Saint Georges (Unknown)
Responsible Party: Sponsor
Other Study IDs: PERCECOVAC
Record Dates: First submitted 2021-05-20; First posted 2021-05-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: vaccination perception
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interview — Face to face semi-directed interviews about perceptions, representations and experiences of Covid-19 vaccination, including six opened-questions

SUMMARY:
SARS COV2, the virus that causes COVID-19, was first described in Wuhan, China. For this pathology, which causes severe respiratory infections, preventing the transmission of the virus has become fundamental, that is why vaccines have been developed. In France, this vaccination campaign took place in a context where the lack of confidence in vaccination is high:

According to a November 2020 IFOP poll, only 41% of French respondents were willing to be vaccinated against COVID-19.

To our knowledge, there are still few qualitative studies on vaccination on the current issue of vaccination against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patient with a scheduled appointment in consultation or at the vaccination centre
* Not opposed to participation in the protocol

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient unable to give free and informed consent
* Patient under court protection
* Patient without the cognitive capacity to ensure an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without comorbidities consulting the Villeneuve Saint Georges Hospital for COVID-19 vaccination or for a scheduled consultation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Perceptions, representations and experiences of Covid-19 vaccination | 1 hour
  Interview based on 6 opened questions

SECONDARY OUTCOMES:
Key elements to improve the medical discourse on vaccination | 1 hour
  Interview based on 6 opened questions

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Villeneuve-Saint-Georges, Villeneuve-Saint-Georges, France

IPD SHARING:
Plan to Share IPD: No